CLINICAL TRIAL: NCT00010647
Title: Cost-Effectiveness of and Long-Term Outcomes Following Acupuncture Treatment for Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000084-01P1 (NIH); P50AT000084-01 (NIH); NCT00009113 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2004-03-25 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to estimate the cost-effectiveness of acupuncture and to determine the long-term outcomes and health care utilization of people with osteoarthritis (OA) of the knee.

DETAILED DESCRIPTION:
Osteoarthritis (OA) makes up a large proportion of the disability and economic costs in the U.S. The knee is the most common site of OA and is a common cause of disability and the leading indication of total knee replacement in the elderly. There are presently no curative therapies for OA. Recently, increased attention has focused on the use of complementary and alternative medicine (CAM) therapies, such as acupuncture, especially for patients who have failed to respond to more standard therapy. Little is known of the long-term health services utilization and outcomes of patients with knee OA. This study will evaluate the cost effectiveness and overall outcomes of acupuncture for OA treatment.

Participants in this study will be randomly assigned to receive either acupuncture or placebo. Surveys and questionnaires will be used to assess participants. Data will be collected on the short- and long-term utilization of health services as well as on pain and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis (OA)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Marc C. Hochberg, Principal Investigator — University of Maryland Osteoporosis Clinic
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Result] Berman BM, Lao L, Langenberg P, Lee WL, Gilpin AM, Hochberg MC. Effectiveness of acupuncture as adjunctive therapy in osteoarthritis of the knee: a randomized, controlled trial. Ann Intern Med. 2004 Dec 21;141(12):901-10. doi: 10.7326/0003-4819-141-12-200412210-00006. PMID 15611487